CLINICAL TRIAL: NCT04413981
Title: Evaluation the Preoperative Anxiety Level of the Surgeons
Status: Completed | Type: Observational
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Tuna Şahin, Specialist of Anesthesiology and Reanimation, Adana City Training and Research Hospital
Other Study IDs: 746
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Preoperative Anxiety
Keywords: surgeon; cortisol; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — salivary cortisol
Oversight: FDA-regulated Drug: No

SUMMARY:
Many studies are present about the preoperative anxiety among patients. But the preoperative anxiety of the surgeons is not studied yet. The aim of this study is to evaluate the preoperative anxiety of the surgeons.100 surgeons consisted of performing operations in general surgery, obstetric and gynecology , orthopedic surgery ,ophthalmology, otorhinolaryngology, plastic and reconstructive surgery, urology, gynecologic oncology, surgical oncology, cardiovascular surgery, pediatric surgery and neurosurgery will be participated in the study. Surgeons will be chosen from the specialist doctor, assistant doctor, doctor lecturer, associate professor and professors.15 minutes prior to the first elective operation of the day, salivary cortisol samples will be taken from the surgeons and they will be asked to fill the evaluation form and State-Trait Anxiety Inventory Form (STAI).

DETAILED DESCRIPTION:
100 surgeons between the ages of 25-55 years will be participated in the study. Surgeons will be consisted of performing operations in general surgery, obstetric and gynecology, orthopedic surgery, ophthalmology, otorhinolaryngology, plastic and reconstructive surgery, urology, gynecologic oncology, surgical oncology, cardiovascular surgery, pediatric surgery and neurosurgery.They will be chosen from the specialist doctor, assistant doctor, doctor lecturer, associate professor and professors. Oral and written informed consent will be obtained from the surgeons.15 minutes prior to the first elective operation of the day salivary cortisol samples will be taken from the surgeons and they will be asked to fill the evaluation form and State-Trait Anxiety Inventory Form (STAI). The evaluation form will include the age, gender of the surgeon, surgical department, academic superscription, years of clinical experience in medical sciences and professions and the name of the surgery which is going to be done.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate the study
* Surgeons planning first elective operation of the day
* 25-55 years

Exclusion Criteria:

* Non volunteers
* Neurological and psychological disorders
* History of anxiolytic , antidepressant drug usage

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Surgeons will be consisted of performing operations in general surgery, obstetric and gynecology, orthopedic surgery, ophtalmology, otorhinolaryngology, plastic and reconstructive surgery, urology, gynecologic oncology, surgical oncology, cardiovascular surgery, pediatric surgery and neurosurgery.They will be chosen from the specialist doctor, assistant doctor, doctor lecturer, associate professor and professors.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
State Trait Anxiety Inventory (STAI) | up to 15 minutes
  State Trait Anxiety Inventory (STAI) form
Serum cortisol sample | up to 5 minutes
  Samples will be taken 15 minutes prior to the first elective surgery of the day

CONTACTS AND LOCATIONS:
Overall Officials: Tuna Şahin, Principal Investigator — Adana City Training and Research Hospital
Locations (1):
- Tuna Şahin, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No